CLINICAL TRIAL: NCT02823210
Title: Clinical and Therapeutic Impact of Molecular Markers in Myeloproliferative Neoplasms (CTIM3)
Brief Title: Clinical and Therapeutic Impact of Molecular Markers in Myeloproliferative Disorders
Acronym: CTIM3
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: TRANSLA13-140
Record Dates: First submitted 2016-06-30; First posted 2016-07-06 (Estimated); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Myeloproliferative Neoplasms
MeSH Terms: conditions — Myeloproliferative Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Molecular markers include mutations in JAK2, MPL, TET2, LNK, CBL, IDH1/2, DNMT3A, EZH2, ASXL1, SF3B1, SRSF2, NRAS/KRAS, and TP53
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Myeloproliferative neoplasms (MPN) are clonal hematopoietic disorders sharing a common natural evolution: a chronic phase, characterized by a major risk of vascular events, followed by an accelerated phase eventually leading to transformation to acute leukemia. MPN include polycythemia vera, essential thrombocythemia, primary myelofibrosis, and rarer entities. During the past years, CML became a paradigm for targeted therapy and personalized cancer medicine. For other MPNs, the discovery of the JAK2V617F mutation followed by many other mutations, opened similar perspectives. However, several questions remain to be answered in MPNs regarding the clinical implication of these major scientific discoveries: what is the clinical impact of JAK2V617F and other molecular biomarkers on the risks of complications and progression? Can these new biomarkers be used in the perspective of a personalized therapy of MPNs? his project will focus on the qualification of a series of known mutations as biomarkers in MPNs based on large multicenter cohorts of patients with well-annotated samples

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from Myeloproliferative neoplasms (MPN) diagnosed between 2005 and 2013
* Sample DNA diagnostics available: 500 mcg
* Untreated or treated with hydroxyurea, ruxolitinib, alpha interferon,
* Patient has given his(her) own consent for the use of the sample for research on the pathology and genetic analyzes

Exclusion Criteria:

* Refused to participate
* Patient treated with another molecule that hydroxyurea, ruxolitinib, or alpha interferon

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Philadelphia-negative Myeloproliferative neoplasms (MPN)
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2016-06; Primary Completion 2019-06 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
cumulative incidence or progression | inclusion

SECONDARY OUTCOMES:
Disease phenotype according to WHO classification | 3 years
  polycythemia vera, essential thrombocythemia, primary myelofibrosis, and others
Treatment response/resistance | 3 years
Mean life-years gained | 3 years
  The analysis will take into consideration the cost of testing, but also the costs of different treatment options with or without testing, and other disease-related costs dependent on treatment
Quality-adjusted life years gained | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Centre d'Investigations Cliniques, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided